CLINICAL TRIAL: NCT00344136
Title: Health Disparities and CVD: Admixture Mapping in the Jackson Heart Study
Brief Title: Identifying Genes That May Increase the Risk for Heart Disease in African Americans
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1344; R01HL084107-01 (NIH)
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Last update posted 2016-07-29 (Estimated); Status verified 2006-10

CONDITIONS: Heart Diseases
Keywords: Blood Pressure, High; Stroke; Hypertension; Diabetes Mellitus; Obesity; Cerebrovascular Accident; Atherosclerosis
MeSH Terms: conditions — Heart Diseases; Hypertension; Stroke; Diabetes Mellitus; Obesity; Atherosclerosis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Heart disease and stroke disproportionately affect African Americans in the United States. These conditions are likely caused by both environmental and genetic factors. This study will attempt to identify specific genes of African and European ancestral origins that may influence the development of heart disease in African Americans.

DETAILED DESCRIPTION:
African Americans have a high risk of developing heart disease and stroke, and are more likely to die from heart-related illnesses than other racial and ethnic groups. A large majority of African Americans are descendants of both African and European ancestors who mixed five to six generations ago. Because only a few generations have passed since that time, it is still possible to identify specific genes, the basic units of heredity, as being either African or European in origin. This is a sub study of the Jackson Heart Study, which is examining the environmental and genetic factors that influence the development of heart disease in African Americans. In this study, researchers will examine genes from participants in the Jackson Heart Study to identify specific African and European genes that influence the development of heart disease in African American men and women.

This study will use genetic samples from individuals participating in the Jackson Heart Study. There will be no study visits for participants. Study researchers will examine the genetic samples and identify specific African and European genes that may influence the development of heart disease, high blood pressure, lipid disorders, left ventricular hypertrophy, and low birth weight.

ELIGIBILITY:
Inclusion Criteria:

* Unrelated African Americans living in Hinds, Rankin, or Madison County, Mississippi enrolled in the Jackson Heart Study

Ages: 21 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5302
Dates: Start 2000-09; Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James G. Wilson, MD, Principal Investigator — University of Mississippi Medical Center and VA Medical Center, Jackson, MS
Locations (1):
- University of Mississippi School of Medicine, Jackson, Mississippi, United States

REFERENCES:
- [Background] Wilson JG, Rotimi CN, Ekunwe L, Royal CD, Crump ME, Wyatt SB, Steffes MW, Adeyemo A, Zhou J, Taylor HA Jr, Jaquish C. Study design for genetic analysis in the Jackson Heart Study. Ethn Dis. 2005 Autumn;15(4 Suppl 6):S6-30-37. PMID 16317983
- [Background] Patterson N, Hattangadi N, Lane B, Lohmueller KE, Hafler DA, Oksenberg JR, Hauser SL, Smith MW, O'Brien SJ, Altshuler D, Daly MJ, Reich D. Methods for high-density admixture mapping of disease genes. Am J Hum Genet. 2004 May;74(5):979-1000. doi: 10.1086/420871. Epub 2004 Apr 14. PMID 15088269